CLINICAL TRIAL: NCT06567210
Title: A Delayed-start Randomized Controlled Trial Comparing the Effects of Online Therapist-guided Cognitive Behavioural and Circadian Therapy for Insomnia Versus Control on Overnight Emotion Regulation and Mental Health Outcomes
Brief Title: The Effects of Insomnia Treatment on Overnight Regulation of Emotional Memories and Risk for Mental Disorders
Acronym: Restless
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14308; 227100/Z/23/Z (Other Grant/Funding Number: Wellcome Trust); GNT1196636 (Other Grant/Funding Number: National Health and Medical Research Council)
Record Dates: First submitted 2024-07-18; First posted 2024-08-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Insomnia Chronic; Anxiety
Keywords: insomnia; anxiety; online cognitive behavioral and circadian therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Delayed-start randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Researchers responsible for randomization and data-analysis will be blinded to the study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate CBCTi (Experimental): Immediate 8-weeks online therapist-guided CBCTi including weekly online modules. Guidance is provided via scheduled and ad hoc communications (e.g., email, messaging, telehealth) between the participant and a clinician/physician
  Interventions: Behavioral: Immediate CBCTi
- Delayed-start control (Other): Participants in the delayed-start control group will not receive any active intervention during two months but will be offered the same therapist-guided CBCTi program thereafter.
  Interventions: Behavioral: Delayed CBCTi

INTERVENTIONS:
Behavioral: Immediate CBCTi — This intervention will be immediately accessible to the CBCTi group. The program is composed of weekly online modules that include written information and interactive components such as schematics, images, videos, and questions. The content of the modules follows traditional and validated cognitive-behavioural therapy for insomnia protocols including sleep education, behavioural strategies (e.g., stimulus control, bedtime retraining, sleep hygiene), cognitive restructuration approaches (e.g., thought reappraisal, imagery, mindfulness), and relaxation practices (progressive muscle relaxation and autogenic training). In addition, further content aims to stabilize and amplify circadian rhythmicity through light exposure in the morning, daytime moderate physical activity, and evening time warm baths. Participants complete daily sleep diaries throughout the intervention.
  Arms: Immediate CBCTi
Behavioral: Delayed CBCTi — This intervention will be accessible after a waiting period of 2 months (i.e, delayed start). The program is composed of weekly online modules that include written information and interactive components such as schematics, images, videos, and questions. The content of the modules follows traditional and validated cognitive-behavioural therapy for insomnia protocols including sleep education, behavioural strategies (e.g., stimulus control, bedtime retraining, sleep hygiene), cognitive restructuration approaches (e.g., thought reappraisal, imagery, mindfulness), and relaxation practices (progressive muscle relaxation and autogenic training). In addition, further content aims to stabilize and amplify circadian rhythmicity through light exposure in the morning, daytime moderate physical activity, and evening time warm baths. Participants complete daily sleep diaries throughout the intervention.
  Arms: Delayed-start control

SUMMARY:
This project aims to elucidate whether CBCTi changes symptom severity or even remission of anxiety disorders as compared with a delayed-start control group. The investigators will use a delayed-start randomized controlled trial in a cohort of individuals with anxiety and insomnia (N=98) to compare the effects of an online therapist-guided cognitive behavioural and circadian therapy for insomnia versus control on overnight emotion regulation and mental health outcomes.

The project will involve at-home assessments and in-lab visits. At-home assessment involves recording sleep and circadian rhythm measures with wearables and daily diaries. Participants will be invited to perform two sleep studies and neuroimaging sessions to investigate the effects of CBCTi on neuroimaging and psychophysiological markers of overnight regulation of emotional distress.

DETAILED DESCRIPTION:
This study is a delayed-start randomized controlled trial comparing the effects of online therapist-guided cognitive behavioural and circadian therapy for insomnia (CBCTi) versus control on emotional regulation and mental health outcomes.

To be enrolled in the study, the participants are required to complete an online prescreening survey followed by a telephone screening interview with further questions and to verbally explain to participants what is required of them in this study. After an interview screening, the participants will receive a finger-pulse oximeter by mail to screen for the presence of obstructive sleep apnoea (3 nights at-home). The device is then returned by pre-paid mail and the recording is analysed to screen for moderate to severe sleep apnoea (oxygen desaturation index ≥ 10). If eligible, the participant will be invited to the Woolcock Institute for a screening visit.

The screening visit starts with a consult with a clinician/physician who performs a medical screening, explains the study, answers questions and addresses concerns, and obtains written informed consent. At the end of the consult, all eligibility criteria have been evaluated and eligible participants are assigned a randomization number i.e., allocated to either the immediate CBCTi-arm or the delayed-start control-arm. The treatment arm consists of an online therapist-guided CBCTi intervention which comprises online sessions to be completed in 8 weeks. Participants in the delayed-start control arm in this study will not receive any active intervention during the first two months but will be offered the same therapist-guided CBCTi program thereafter

During the screening visit, participants will be asked to perform in an audio-visual recording while singing along to "Waltzing Matilda" (karaoke style) and asked to give keywords that relate to at least five negative distressing experiences and an equal number of neutral experiences from the same period. The recording and the keywords will be used to derive the stimuli that are used in the functional MRI tasks (Pre-Post CBCTi). The screening visit is concluded with a demonstration on how to collect data at-home.

Both groups will be asked to perform a week of at-home assessment during 4 timepoints: T0 (baseline), T1 (2 months post-baseline), T2 (4 months post-baseline) and T3 (12 months post-baseline). During the week of at-home assessments, the participants complete questionnaires, keep a sleep diary, and wear an actigraphy-watch, and light and temperature sensor (across 7 days). They are also asked to complete at least four overnight polysomnographic recordings using an EEG headband. At Pre and Post-CBCTi only, they also complete a salivary melatonin collection protocol.

At Pre and Post-CBCTi (i.e., T0 and T1 for immediate group - T1 and T2 for delayed group) , participants are invited to Macquarie University/Woolcock Institute to undergo overnight sleep studies and neuroimaging sessions.

The CBCTi program will be given online via secure platforms and recruitment will primarily be through social media advertisements. The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Macquarie Park, New South Wales, 2109, Australia.

ELIGIBILITY:
Inclusion Criteria:

* (A or B) and (C) A. Diagnosis of insomnia disorder (DSM-5-TR) B. Insomnia Severity Index (ISI) score ≥ 10 C. Generalized Anxiety Disorder (GAD-7) score ≥ 10
* All sexes and genders.
* Between 18 and 45 years of age.
* Able to provide informed consent.
* Proficient in English.

Exclusion Criteria:

x Sleep or circadian disorder other than insomnia (e.g., hypersomnolence, periodic limb movement disorder, advanced or delayed sleep phase disorder, moderate to severe sleep apnoea disorder based on previous sleep study with an apnea-hypopnea index ≥ 15 and/or finger-pulse oximetry oxygen desaturation index (ODI) ≥ 10).

* Current or history of neurological disorders (e.g., stroke, brain injury).
* Current or history of bipolar disorder, psychosis, or moderate to severe obsessive-compulsive disorder.
* Current uncontrolled mental health disorders requiring specialist care, other than major depression and anxiety disorders.
* Centrally active agents or presence of medical condition that may affect participation.
* Pregnancy or actively trying to conceive, or lactating.
* Shift work for at least 2 shifts per week in the past 3 months (i.e., work between 21:00 and 6:00).
* Travel across time zones over 3 hours difference in the previous 30 days (will require a 1-day adjustment period per hour of time zone travelled).
* Unwilling to know about potential incidental findings.
* No consent or adherence to instructions for any part of the study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) score | 2 months, 4 months, 12 months
  Self-report measures of anxiety symptoms and severity. GAD-7 consists of 7 Likert-scale questions with a total score ranging from 0 to 21 (with higher scores indicating more severe anxiety)
Anxiety Disorder diagnosis | 2 months, 4 months, 12 months
  Clinician-diagnosed anxiety disorder in accordance with the DSM-5-TR using the Mini-International Neuropsychiatric Interview

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) score | 2 months, 4 months, 12 months
  Self-report measures of insomnia symptoms and severity. ISI consists of 7 Likert-scale questions with a total score ranging from 0 to 28 (with higher scores indicating more severe insomnia)
EEG sleep efficiency (SE - %) | 2 months, 4 months, 12 months
  Mean SE derived from at-home sleep recordings (total sleep time/time in bed*100)
EEG total sleep time (TST - minutes) | 2 months, 4 months, 12 months
  Mean TST derived from at-home sleep recordings
EEG wake duration (minutes) | 2 months, 4 months, 12 months
  Mean wake after sleep onset (WASO) derived from at-home sleep recordings
EEG sleep onset latency (SOL - minutes) | 2 months, 4 months, 12 months
  Mean SOL derived from at-home sleep recordings
EEG sleep stages (%) | 2 months, 4 months, 12 months
  Mean time spent in sleep stages (per total sleep period) derived from at-home sleep recordings
Actigraphy sleep efficiency (%) | 2 months, 4 months, 12 months
  Mean SE derived from actigraphy recording (total sleep time/time in bed*100)
Actigraphy total sleep duration (minutes) | 2 months, 4 months, 12 months
  Mean TST derived from actigraphy recordings
Actigraphy wake duration (minutes) | 2 months, 4 months, 12 months
  Mean WASO derived from actigraphy recordings
Actigraphy sleep onset latency (minutes) | 2 months, 4 months, 12 months
  Mean SOL derived from actigraphy recordings
7-days light exposure (lux) | 2 months, 4 months, 12 months
  derived from at-home continuous light recording during the day
Hour of Dim-Light Melatonin Onset (HDLMO - hour) | 2 months
  derived from at-home collection of saliva samples
3-days distal-proximal skin-temperature gradients (DPG) | 2 months, 4 months, 12 months
  derived from at-home collection of continuous skin temperature (4 locations)
Self-reported sleep duration (min) | 2 months, 4 months, 12 months
  Mean TST derived from sleep diaries
Self-reported wake duration (min) | 2 months, 4 months, 12 months
  Mean WASO derived from sleep diaries
Self-reported sleep onset latency (min) | 2 months, 4 months, 12 months
  Mean SOL derived from sleep diaries
Self-reported sleep quality (out of 5) | 2 months, 4 months, 12 months
  Mean sleep quality derived from sleep diaries on a scale from 0 to 4 (very poor sleep to very good sleep)
Sleep misperception index (SPI - %) | 2 months, 4 months, 12 months
  SPI derived from subjective TST and objective TST (Subj/Obj*100)

OTHER OUTCOMES:
Sleep electroencephalographic (EEG) spectral power | 2 months
  derived from polysomnographic (PSG) recordings in-lab: absolute and relative spectral power for band frequencies: slow oscillations (0.25-1.25Hz), delta (0.25-4Hz), theta (4.25-8Hz), alpha (8.25-11.75Hz), sigma (12-16Hz), low beta (16.25-19Hz), high beta (19.25-35Hz) for all stages.
Sleep electroencephalographic (EEG) neuro-oscillatory coupling | 2 months
  derived from PSG recordings in-lab - phase-amplitude coupling measures (modulation index, preferred phase)
Functional connectivity patterns in resting-state brain networks | 2 months
  measured by network-wise dual-regression independent component analysis (FMRIB FSL) with the whole-brain voxel-wise connectivity strength is the dependent variable
EEG sleep-related brain oscillations (characteristics) | 2 months
  EEG neurophysiological events derived from PSG recordings in-lab : density, duration, peak frequency, amplitude, number
Brain activation during tasks using functional magnetic resonance imaging | 2 months
  Whole-brain voxel-wise brain activation maps of the blood-oxygen dependent signal response to emotional stimuli during the Karaoke and Autobiography tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Wassing, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
All study team members have access to the dataset. Other Woolcock-affiliated staff may also request access to the non-identifiable dataset, which will be considered by the principal investigator and co-investigators. A copy of the non-identifiable dataset may be requested by academic collaborators not affiliated with the Woolcock through a data request form, which outlines the investigators, aims and hypotheses, data to be included, a statistical analysis plan, ethics approval, and security measures.

REFERENCES:
- [Background] Hertenstein E, Feige B, Gmeiner T, Kienzler C, Spiegelhalder K, Johann A, Jansson-Frojmark M, Palagini L, Rucker G, Riemann D, Baglioni C. Insomnia as a predictor of mental disorders: A systematic review and meta-analysis. Sleep Med Rev. 2019 Feb;43:96-105. doi: 10.1016/j.smrv.2018.10.006. Epub 2018 Nov 16. PMID 30537570
- [Background] Taylor DJ, Pruiksma KE. Cognitive and behavioural therapy for insomnia (CBT-I) in psychiatric populations: a systematic review. Int Rev Psychiatry. 2014 Apr;26(2):205-13. doi: 10.3109/09540261.2014.902808. PMID 24892895
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] Leerssen J, Lakbila-Kamal O, Dekkers LMS, Ikelaar SLC, Albers ACW, Blanken TF, Lancee J, van der Lande GJM, Maksimovic T, Mastenbroek SE, Reesen JE, van de Ven S, van der Zweerde T, Foster-Dingley JC, Van Someren EJW. Treating Insomnia with High Risk of Depression Using Therapist-Guided Digital Cognitive, Behavioral, and Circadian Rhythm Support Interventions to Prevent Worsening of Depressive Symptoms: A Randomized Controlled Trial. Psychother Psychosom. 2022;91(3):168-179. doi: 10.1159/000520282. Epub 2021 Dec 6. PMID 34872087
- [Background] Christensen H, Batterham PJ, Gosling JA, Ritterband LM, Griffiths KM, Thorndike FP, Glozier N, O'Dea B, Hickie IB, Mackinnon AJ. Effectiveness of an online insomnia program (SHUTi) for prevention of depressive episodes (the GoodNight Study): a randomised controlled trial. Lancet Psychiatry. 2016 Apr;3(4):333-41. doi: 10.1016/S2215-0366(15)00536-2. Epub 2016 Jan 28. PMID 26827250
- [Background] Wassing R, Lakbila-Kamal O, Ramautar JR, Stoffers D, Schalkwijk F, Van Someren EJW. Restless REM Sleep Impedes Overnight Amygdala Adaptation. Curr Biol. 2019 Jul 22;29(14):2351-2358.e4. doi: 10.1016/j.cub.2019.06.034. Epub 2019 Jul 11. PMID 31303489
- [Background] Wassing R, Schalkwijk F, Lakbila-Kamal O, Ramautar JR, Stoffers D, Mutsaerts HJMM, Talamini LM, Van Someren EJW. Haunted by the past: old emotions remain salient in insomnia disorder. Brain. 2019 Jun 1;142(6):1783-1796. doi: 10.1093/brain/awz089. PMID 31135050
- [Background] Lancee J, van Straten A, Morina N, Kaldo V, Kamphuis JH. Guided Online or Face-to-Face Cognitive Behavioral Treatment for Insomnia: A Randomized Wait-List Controlled Trial. Sleep. 2016 Jan 1;39(1):183-91. doi: 10.5665/sleep.5344. PMID 26414893
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Berntsen D, Hoyle RH, Rubin DC. The Autobiographical Recollection Test (ART): A Measure of Individual Differences in Autobiographical Memory. J Appl Res Mem Cogn. 2019 Sep;8(3):305-318. doi: 10.1016/j.jarmac.2019.06.005. Epub 2019 Jul 26. PMID 31700775